CLINICAL TRIAL: NCT05917119
Title: Bright Light Therapy for Residual Daytime Symptoms Associated With Obstructive Sleep Apnea
Brief Title: Bright Light Therapy for OSA
Acronym: BrightDaysII
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: F4531-R
Record Dates: First submitted 2023-06-14; First posted 2023-06-23 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Obstructive Sleep Apnea
Keywords: Obstructive sleep apnea; CPAP; Residual daytime sleepiness; Depressive symptoms
MeSH Terms: conditions — Sleep Apnea, Obstructive; Depression

STUDY DESIGN:
Intervention Model Description: single blind crossover design with randomized condition order
Who Masked: Participant
Masking Description: Participants are not told which arm is active versus sham
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- BLT (Experimental): Bright light therapy delivered via glasses
  Interventions: Other: BLT
- s-BLT (Sham Comparator): Sham Bright light therapy
  Interventions: Other: s-BLT

INTERVENTIONS:
Other: BLT — Bright light therapy delivered via glasses
  Other Names: Bright light therapy-Active intervention
  Arms: BLT
Other: s-BLT — sham delivered with bright light therapy glasses to which a neutral density filter has been applied
  Other Names: sham-Bright light therapy
  Arms: s-BLT

SUMMARY:
Persistent daytime symptoms of sleepiness in individuals with obstructive sleep apnea (OSA) who are using Continuous Positive Airway Pressure (CPAP) are associated with adverse long term medical and functional outcomes. Supplementary exposure to bright light has beneficial effects on sleep quality and daytime vigilance in healthy individuals and it has been increasingly applied in a variety of sleep and neuropsychiatric conditions. This study will explore the role of Bright Light Therapy (BLT), a well-established non-pharmacological intervention for circadian disturbances, for the treatment of residual daytime symptoms of OSA which do not respond to CPAP. BLT will be delivered via therapy glasses in a cross-over design, where each participant will be exposed to active treatment and sham treatment (4 weeks in each arm) in a randomized order. The hypothesis is that participants will demonstrate improvements in the variables of interest during the four-week active treatment portion of the eight-week crossover study, compared to the four-week sham treatment portion.

DETAILED DESCRIPTION:
Persistent daytime symptoms of sleepiness in individuals with obstructive sleep apnea (OSA) who are using Continuous Positive Airway Pressure (CPAP) are associated with adverse long term medical and functional outcomes. Supplementary exposure to bright light has beneficial effects on sleep quality and daytime vigilance in healthy individuals and it has been increasingly applied in a variety of sleep and neuropsychiatric conditions. This study will explore the role of Bright Light Therapy (BLT), a well-established non-pharmacological intervention for circadian disturbances, for the treatment of residual daytime symptoms of OSA which do not respond to CPAP. BLT will be delivered via therapy glasses in a cross-over design, where each participant will be exposed to active treatment and sham treatment (4 weeks in each arm) in a randomized order. The hypothesis is that participants will demonstrate improvements in the variables of interest during the four-week active treatment portion of the eight-week crossover study, compared to the four-week sham treatment portion.

ELIGIBILITY:
Inclusion Criteria:

* Documented diagnosis of OSA
* Currently on CPAP or BiPAP for at least 3 months

  * with documented adherence (defined as wearing CPAP/BiPAP for >6h/night on at least 75% of nights), and adequate control of sleep apnea, as indicated by an AHI of 10 or less when on CPAP
* Excessive residual daytime sleepiness (Epworth score > 10)
* If taking alertness promoting medication, the investigators will require that they are on a stable dose for at least one month prior to entering the study and that they refrain from dose changes while participating in the study
* If already prescribed BLT, subjects must not have used it for at least one month prior to participating

Exclusion Criteria:

* Shift work
* Travel across time zones in the past month
* Narcolepsy
* Regular hypnotics use
* Decompensated congestive heart failure (CHF)
* Primary central sleep apnea, needing O2 therapy via nasal cannula
* Poorly controlled diabetes (HgA1c>8%)
* Active substance use disorder
* Dementia
* Untreated bipolar disorder

  * the investigators will consider individuals with a diagnosis of bipolar disorder who are currently in treatment and stable
* Macular degeneration, recent lasik surgery (within 3 months)
* Legally blind
* Taking medication that will cause photosensitivity to blue-green light spectrum wavelength
* Already using bright light therapy

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-10-26 (Actual); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Epworth sleepiness scale | baseline, week 4 (end of treatment 1), week 8 (end of wash out), week 12 (end of treatment 2)
  self report questionnaire assessing daytime drowsiness and tendency to fall asleep if inactive
Change in QIDS score | baseline, week 4 (end of treatment 1), week 8 (end of wash out), week 12 (end of treatment 2)
  self report assessment of depressive symptoms severity

CONTACTS AND LOCATIONS:
Overall Officials: Isabella Soreca, MD, Principal Investigator — VA Pittsburgh Healthcare System University Drive Division, Pittsburgh, PA
Locations (1):
- VA Pittsburgh Healthcare System University Drive Division, Pittsburgh, PA, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No